CLINICAL TRIAL: NCT04246476
Title: Sing for Your Saunter: Using Self-generated Rhythmic Cues to Enhance Gait in Parkinson's
Brief Title: Sing for Your Saunter
Acronym: SFYS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Gammon M Earhart, Director, Program in Physical Therapy, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201908117; 1R61AT010753-01 (NIH)
Record Dates: First submitted 2020-01-24; First posted 2020-01-29 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease
Keywords: parkinson disease; music; imaging; mental singing; gait
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self cueing (Experimental): People living with Parkinson disease and controls walking with self-generated rhythmic cues.
  Interventions: Behavioral: Mentally singing; Behavioral: Listening to music
- External cueing (Active Comparator): People living with Parkinson disease and controls walking to external rhythmic cues (i.e., music).
  Interventions: Behavioral: Mentally singing; Behavioral: Listening to music

INTERVENTIONS:
Behavioral: Mentally singing — All participants (people with PD and age-matched controls) sing their song in their head and match their footfalls or finger tapping to the beat.
Behavioral: Listening to music — All participants (people with PD and age-matched controls) listen to their song and match their footfalls or finger tapping to the beat.

SUMMARY:
Older adults, and particularly those with Parkinson disease (PD), may experience walking difficulties that negatively impact their daily function and quality of life. This project will examine the impact of music and mentally singing on walking performance, with a goal of understanding what types of rhythmic cues are most helpful. Our pilot work suggests that imagined, mental singing (i.e., singing in your head) while while walking helps people walk faster with greater stability, whereas walking to music also helps people walk faster but with reduced stability.

In Aim 1, the investigators will compare walking while mentally singing to walking while listening to music, using personalized cues tailored to each person's walking performance. The investigators hypothesize stride time variability will be less in the mental singing condition compared to listening to music; and that mental singing and listening to music will improve gait speed similarly as compared to the uncued condition. The investigators will also test whether finger tapping, a rhythmic task similar to walking in many ways, responds similarly while mentally singing and listening to music.

In Aim 2, the investigator will investigate the brain mechanisms underlying the enhancements in movement performance seen with mental signing or listening to music. The investigators will use magnetic resonance imaging (MRI) to measure brain activity during finger tapping with and without various cues to understand which areas of the brain are more or less responsive to the cues. The investigators hypothesize individuals with PD will exhibit lesser activation of putamen and greater activation of cortical motor areas and cerebellum compared to controls in all tapping conditions; and internal, mental singing during tapping will elicit greater activation of the putamen and lesser activation of cortical motor areas in both groups compared to uncued tapping and tapping while listening to music.

DETAILED DESCRIPTION:
During this observational study, all participants will attend two visits 4-10 days apart. At the first visit, all participants (participants with PD and age-matched controls) will wear wearable sensors during the following tasks: walking with no cues; walking while listening to music; and walking while mentally singing. The wearable sensors will measure gait parameters including gait speed and stride time variability. All participants will also conduct the following tasks while finger tapping on a keyboard: tapping with no cues; tapping while listening to music; and tapping while mentally singing.

At the second visit, all participants (participants with PD and age-matched controls) will perform the following tasks during imaging: uncued tapping; listening to music (no tapping); mentally singing (no tapping); listening to music and tapping; and mentally singing and tapping.

ELIGIBILITY:
Inclusion Criteria for all participants:

* at least 30 years of age;
* willing and able to provide informed consent;
* right-handed or ambidextrous;
* normal hearing;
* weight less than 250 lbs; and
* able to walk for 10 continuous minutes independently.

Inclusion criteria for participants with PD also include:

* diagnosis of idiopathic, typical Parkinson disease according to the United Kingdom Brain Bank Criteria;
* Hoehn & Yahr stages 2-3 (mild to moderate disease severity);
* stable on all PD medications for at least 2 months prior to study entry;
* a score of 1 or less on item # 7 on the New Freezing of Gait Questionnaire; and
* score of ≥ 1 on the Movement Disorder Society - Unified Parkinson Disease Rating Scale (MDS-UPDRS)-III Item #10 indicating observable gait impairment.

Exclusion Criteria for both groups include:

* diagnosis of any other neurological condition;
* significant cognitive impairment;
* unstable medical or concomitant illnesses or psychiatric conditions which, in the opinion of the investigators, would preclude successful participation;
* cardiac problems that interfere with ability to safely participate (i.e., uncontrolled congestive heart failure, myocardial infarction in past 6 months, complex cardiac arrhythmias, significant left ventricular dysfunction, dyspnea on exertion, chest pain or pressure, resting tachycardia (>100 beats/min); uncontrolled BP (resting systolic BP >160 mmHg or diastolic BP >100 mmHg));
* orthopedic problems in the lower extremities or spine that may limit walking (i.e., severe arthritis, spinal stenosis);
* contraindications for magnetic resonance imaging (e.g., metallic implants); or
* uncontrolled tremor or dyskinesia (while on PD medications if applicable).

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gammon Earhart, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine Program in Physical Therapy, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants in both groups completed all conditions (i.e., uncued, mental singing and music) at all tempos (i.e., 90, 100, 110 and 120% of baseline uncued cadence).
Groups:
- Parkinson Disease Group: People living with Parkinson disease
- Healthy Controls: Healthy controls age-matched to Parkinson disease group
Period: Overall Study
Arm/Group | Parkinson Disease Group | Healthy Controls
Started | 29 | 29
Completed | 29 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Reporting results separately for group with PD and healthy controls, though both groups were assigned to same walking conditions
Groups:
- Parkinson Group: People living with Parkinson disease walking with and without rhythmic cues.
  Mentally singing: All participants (people with PD and age-matched controls) sing their song in their head and match their footfalls or finger tapping to the beat.
  Music: All participants (people with PD and age-matched controls) listen to their song and match their footfalls or finger tapping to the beat.
  Uncued: no music and no singing
- Healthy Control Group: Healthy controls walking with and without rhythmic cues.
  Mentally singing: All participants (people with PD and age-matched controls) sing their song in their head and match their footfalls or finger tapping to the beat.
  Music: All participants (people with PD and age-matched controls) listen to their song and match their footfalls or finger tapping to the beat.
  Uncued: no music and no singing
- Total: Total of all reporting groups
Arm/Group | Parkinson Group | Healthy Control Group | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 13 | 25
  >=65 years | 17 | 16 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 14 | 14 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 28 | 28 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Mini Mental Status Exam [Median (Full Range); unit: units on a scale] — Scores on the Mini Mental Status range from 0 to 30, with higher scores indicating better cognitive function. Scores below 26 indicate cognitive impairment.
  units on a scale | 29 [27 to 30] | 29 [26 to 30] | 29 [26 to 30]

OUTCOME MEASURES:

1. Primary Outcome: Gait Speed
Description: Measured with wearable sensors by APDM Wearable Technology
Time Frame: Baseline
Population: Results are presented separately for each group and for each cueing condition (uncued, music or mental singing) and tempo (90, 100, 110, 120%).
Measure: Mean (Standard Deviation); unit: meters per second
Groups:
- Parkinson Disease Group: People with Parkinson disease
- Healthy Controls: Healthy controls age-matched to the Parkinson disease group
Arm/Group | Parkinson Disease Group | Healthy Controls
Number analyzed (Participants) | 29 | 29
meters per second
  Uncued | 1.12 (.16) | 1.17 (.13)
  Music 90% | 1.04 (.15) | 1.09 (.15)
  Mental singing 90% | 1.16 (.16) | 1.11 (.13)
  Music 100% | 1.13 (.16) | 1.17 (.15)
  Mental singing 100% | 1.13 (.17) | 1.19 (.15)
  Music 110% | 1.22 (.19) | 1.24 (.16)
  Mental singing 110% | 1.21 (.17) | 1.23 (.16)
  Music 120% | 1.29 (.2) | 1.31 (.17)
  Mental singing 120% | 1.27 (.17) | 1.29 (.15)

2. Primary Outcome: Stride Length Variability
Description: Measured with wearable sensors by APDM Wearable Technology
Time Frame: Baseline
Population: Results are presented separately for each group in each condition (uncued, music, mental singing) at each tempo (90, 100, 110, 120% of uncued).
Measure: Mean (Standard Deviation); unit: coefficient of variation
Groups:
- Parkinson Disease Gruop: People with Parkinson disease
Arm/Group | Parkinson Disease Gruop | Healthy Controls
Number analyzed (Participants) | 29 | 29
coefficient of variation
  Uncued | .014 (.003) | .013 (.005)
  Music 90% | .015 (.005) | .014 (.003)
  Mental singing 90% | .013 (.006) | .012 (.003)
  Music 100% | .013 (.005) | .014 (.004)
  Mental singing 100% | .013 (.005) | .011 (.002)
  Music 110% | .014 (.009) | .014 (.004)
  Mental singing 110% | .012 (.007) | .012 (.003)
  Music 120% | .016 (.009) | .014 (.006)
  Mental singing 120% | .012 (.005) | .011 (.005)

3. Secondary Outcome: Brain Activity (BOLD Signal)
Description: We analyzed the Blood Oxygen Level Dependent (BOLD) signal in the brain to determine where there were areas of significant changes in brain activity, relative to rest, when participants were moving with no cue (uncued), moving to the beat during self cueing (mental singing) and moving to the best during external cueing (music). BOLD values are reported are Beta weights. Positive values indicate an increase in activity relative to rest and negative values indicate a decrease in activity relative to rest.
Time Frame: Baseline
Population: Results are presented separately for each group in each condition (uncued, music, mental singing).
Measure: Mean (Standard Deviation); unit: Beta weights (arbitrary units)
Arm/Group | Parkinson Disease Group | Healthy Controls
Number analyzed (Participants) | 27 | 28
Beta weights (arbitrary units)
  Uncued Left Putamen | -.054 (.217) | -.017 (.189)
  Uncued Right Putamen | -.053 (.181) | -.053 (.143)
  Uncued Bilateral Primary Somatosensory Cortex | .069 (.260) | .139 (.221)
  Music Left Putamen | -.027 (.268) | .091 (.293)
  Music Right Putamen | -.069 (.199) | .035 (.233)
  Music Bilateral Auditory Cortex | .102 (.240) | .246 (.357)
  Music Bilateral Primary Somatosensory Cortex | .096 (.183) | .218 (.279)
  Mental singing Left Putamen | -.0001 (.272) | .114 (.296)
  Mental Singing Right Putamen | -.063 (.250) | .024 (.279)
  Mental singing Bilateral Primary Somatosensory Cortex | .177 (.291) | .258 (.394)

ADVERSE EVENTS:
Time Frame: Monitoring of participants during two separate visits of a few hours each on 2 different days no more than 2 weeks apart.
Description: Participants were supervised throughout their time in the two sessions so adverse events were monitored continuously
Groups:
- Parkinson Disease Group: Individuals with Parkinson disease
- Healthy Control Group: Healthy controls age-matched to Parkinson disease group
Arm/Group | Parkinson Disease Group | Healthy Control Group
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT04246476/Prot_SAP_000.pdf